CLINICAL TRIAL: NCT03882853
Title: The Effect of Yoga Asana 'Vrksasana (Tree Pose)' on Balance in the Patients With Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, MD, Research Assistant of PMR, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FTR OP
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Osteoporosis
Keywords: yoga; osteoporosis; balance; tree pose; asana
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative exercise group (CEG) (Active Comparator): Conservative exercise group
  Interventions: Other: Conservative exercise group
- Tree pose added exercise group (TPAEG) (Experimental): Tree pose added exercise group
  Interventions: Other: Conservative exercise group; Other: Tree pose added exercise group

INTERVENTIONS:
Other: Conservative exercise group — The group will be thought exercise series which based on recommendations published on October 2016 by UK national osteoporosis foundation.Handouts including pictures and narrations of the exercises will be given to patients. Patients would be encouraged to perform the exercises 5 days a week. A diary will be given to note the days exercises completed.
  Other Names: CEG
Other: Tree pose added exercise group — The group will be thought exercise series which will be based on recommendations which is published on October 2016 by UK national osteoporosis foundation, also be taught "tree pose" of yoga. Handouts including pictures and narrations of the exercises will be given to patients. Patients would be encouraged to perform the exercises 5 days a week. A diary will be given to note the days exercises completed.
  Other Names: TPAEG
  Arms: Tree pose added exercise group (TPAEG)

SUMMARY:
Patients with T score of bone mineral densitometry less than or equal to -2.5 will be included in the study. Initial evaluation consists of obtaining demographic data, performing international physical activity questionnaire (short form) Additionally; Berg balance test, timed sit and walk test, single leg stance test, tandem walk test, tandem stance test will be performed. Baseline static and dynamic balance scores of patients will be determined by the Corebalance Premiere-19 balance device. After acclimation the device and tests, 3 measurements will be made and the most successful score will be taken. The lowest value will be showing best performance. After the first evaluation, patients will be randomized using windows excel randomization option to two groups by another observer. Patients will be blinded about which exercise group they will be separated to. Both groups will be thought exercise series which will be based on recommendations which is published on October 2016 by UK national osteoporosis foundation. Patients would be encouraged to perform the exercises on recommended basis and handouts will be given to patients in both groups. The yoga group will also be taught "tree pose".

Patients will be encouraged to note their exercises regularly on daily basis. Patients will be reevaluated after first and third months and balance tests will be re-performed to determine the effect of given exercises.

Exclusion criteria

* Neurological or vestibule dysfunctions which may affect balance
* Severe mental disturbances effecting communication
* Locomotor dysfunction which prevents patient to perform balance tests
* Active musculoskeletal pathology which disrupt performing exercises.

DETAILED DESCRIPTION:
Patients with osteoporosis who applied to PMR outpatient clinic of Istanbul Medeniyet University Goztepe Training and Research Hospital will be included in the study. Informed consent detailing the purpose and content of the study will be obtained from patients. Initial evaluation of patients will be performed by the same doctor. Initial evaluation consists of obtaining demographic data and performing international physical activity questionnaire (short form) to evaluate physical activity frequencies of patients. Additionally; Berg balance test, timed sit and walk test, single leg stance test, tandem walk test, tandem stance test will be performed. Baseline static and dynamic balance scores of patients will be determined by the Corebalance Premiere-19 balance device. After acclimation the device and tests, 3 measurements will be made and the most successful score will be taken. The lowest value will be showing best performance. After the first evaluation, patients will be randomized using windows excel randomization option to two groups by another observer. Patients will be blinded about which exercise group they will be separated to. To learn the exercises the patient will be referred to physiatrist Ozge Solakoglu who completed a 200-hour yoga teacher training programme certificated by Yoga Alliance. Both groups will be thought exercise series which will be based on recommendations which is published on October 2016 by UK national osteoporosis foundation. Patients would be encouraged to perform the exercises on recommended basis and handouts will be given to patients in both groups. The yoga group will also be taught "tree pose".

Patients will be encouraged to note their exercises regularly on daily basis. Patients will be reevaluated after first and third months and balance tests will be re-performed to determine the effect of given exercises.

Inclusion criteria

- Patients with T score of bone mineral densitometry lower than -2.5.-

Exclusion criteria

* Neurological or vestibule dysfunctions which may affect balance
* Severe mental disturbances effecting communication
* Locomotor dysfunction which prevents patient to perform balance tests
* Active musculoskeletal pathology which disrupt performing exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T score of bone mineral densitometry lower than -2.5.

Exclusion Criteria:

* Neurological or vestibule dysfunctions which may affect balance
* Severe mental disturbances effecting communication
* Locomotor dysfunction which prevents patient to perform balance tests
* Active musculoskeletal pathology which disrupt performing exercises.

Ages: 35 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Static balance score | 5 min.
  The Korebalance Premiere-19 device and software will be used to make balance assessment. Static test requires standing steady and balancing on the platform, keeping the cross-hairs of cursor in the center of the test pattern. The score indicates the deviation of user's center of gravity from the center of the pattern. After familirization of the patient to the test, the lowest score of three measurements will be noted. The lowest score gives the most successfull scores of test.

SECONDARY OUTCOMES:
Dynamic balance score | 5 min.
  The Korebalance Premiere-19 device and software will be used to make balance assessment. Dinamic test offers a moving cursor that the user ''follows''. Cursor patterns a clock-wise circle. After familirization of the patient to the test, the lowest score of three measurements will be noted. The lowest score gives the most successfull scores of test.
Berg balance test score | 10 min.
  14-item scale designed to measure balance of the older adult in a clinical setting. A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Total Score is 56. Score of 41-56 indicates low fall risk, 21-40 indicates medium fall risk, 0 -20 indicates high fall risk. It is supported a cut off score of 45/56 for independent safe ambulation.
Timed sit and walk test score | 1 min.
  The objective is to determine fall risk and measure the progress of balance, sit to stand and walking. The patient starts in a seated position, the patient stands up upon command, walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated. The subject is allowed to use an assistive device. If an assistive device is used, it will be documented.
Single leg stance test score | 1 min
  It is used to test the static balance and postural control. It is performed eyes open and arms on the hips. The patient must stand unassisted on one leg. The time between one foot is flexed off the floor to the time when it touches the ground. If less then 30 second, it will be noted, patients stands with more than 30 seconds accepted succesfull.
Tandem walk test score | 1 min
  The patient will asked to walk in a straight line with one foot immediately in front of the other (heel to toe) for 10 footstep for each foot. The time will be documented.
Tandem stance test score | 1 min
  The patient will be ask to stand tandem (heel to toe) for 30 seconds. Lower than 30 second will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Solakoglu, MD, Principal Investigator — Istanbul Medeniyet University Physical Medicine and Rehaiblitation Clinic
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine, Physical Medicine and Rehabilitation Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solakoglu O, Dogruoz Karatekin B, Yumusakhuylu Y, Mesci E, Icagasioglu A. The Effect of Yoga Asana "Vrksasana (Tree Pose)" on Balance in Patients With Postmenopausal Osteoporosis: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Mar 1;101(3):255-261. doi: 10.1097/PHM.0000000000001785. PMID 33990483